CLINICAL TRIAL: NCT01543893
Title: Danish: Integreret Motion på Arbejdspladsen (IRMA) English: Implementation of Exercise at the Workplace
Brief Title: Effect of Personal Versus Video Instruction in Elastic Resistance Exercise on Technical Execution (IRMA05)
Acronym: IRMA05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Lars L. Andersen, Principal Investigator, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRMA05
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Musculoskeletal Disorders
Keywords: neck pain; shoulder pain; resistance training
MeSH Terms: conditions — Musculoskeletal Diseases; Neck Pain; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video instruction (Experimental): Participants will receive an elastic resistance tubing, an internet link and a poster with instructions to perform four different elastic resistance exercises Participants are encouraged to perform the exercises daily on weekdays during the next two weeks
  Link to exercises: http://www.jobogkrop.dk/Ondt-i-muskler-og-led/Ondt-i-nakke-skulder-og-arm/Elastikoevelser-for-nakke-skulder-og-arm
  Interventions: Behavioral: Video instruction
- Personal instruction (Active Comparator): Participants will receive an elastic resistance tubing, an internet link and a poster with instructions to perform four different elastic resistance exercises Participants are encouraged to perform the exercises daily on weekdays during the next two weeks In addition to the video group, this group will also receive personal instruction during the two weeks.
  Link to exercises: http://www.jobogkrop.dk/Ondt-i-muskler-og-led/Ondt-i-nakke-skulder-og-arm/Elastikoevelser-for-nakke-skulder-og-arm
  Interventions: Behavioral: Personal instruction

INTERVENTIONS:
Behavioral: Video instruction — Participants will receive an elastic resistance tubing, an internet link and a poster with instructions to perform four different elastic resistance exercises Participants are encouraged to perform the exercises daily on weekdays during the next two weeks
  Link to exercises: http://www.jobogkrop.dk/Ondt-i-muskler-og-led/Ondt-i-nakke-skulder-og-arm/Elastikoevelser-for-nakke-skulder-og-arm
  Arms: Video instruction
Behavioral: Personal instruction — Participants will receive an elastic resistance tubing, an internet link and a poster with instructions to perform four different elastic resistance exercises Participants are encouraged to perform the exercises daily on weekdays during the next two weeks In addition to the video group, this group will also receive personal instruction during the two weeks.
  Link to exercises: http://www.jobogkrop.dk/Ondt-i-muskler-og-led/Ondt-i-nakke-skulder-og-arm/Elastikoevelser-for-nakke-skulder-og-arm
  Arms: Personal instruction

SUMMARY:
Resistance training is widely used in training and rehabilitation. During recent years elastic resistance training has become increasingly popular for preventing or relieving neck/shoulder/arm pain among sedentary employees. While most research studies documenting positive effects of such interventions have used training instructors, most training in practice does not use an instructor but rather depends on information from other sources such as the internet. Here the investigators examine - in a outcome assessor blinded randomized controlled trial - the effect of 2 weeks elastic resistance training for the neck/shoulder/arm with personal versus video instruction on technical execution.

ELIGIBILITY:
Inclusion Criteria:

* neck or shoulder pain

Exclusion Criteria:

* blood pressure above 160/100 mmHg
* pregnancy
* life-threatening disease

Ages: 18 Years to 67 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Technical execution | 2 weeks after randomization
  * joint positions will be scored for each individual joint and plane on a 5 point scale according to standard execution according to images
  * a total score (primary outcome) will be calculated by summing scores from each individual joint position

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — Professor
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

REFERENCES:
- See also: Company website — http://www.arbejdsmiljoforskning.dk